CLINICAL TRIAL: NCT03451253
Title: Effects of an Amino Acid Mixture Versus a Sugar Based Sports Drink on Gastrointestinal Function, Inflammation and Fluid Balance: A Pilot Study in Patients With Inflammatory Bowel Disease
Brief Title: Effects of an Amino Acid Mixture on Gastrointestinal Function, Inflammation and Fluid Balance: A Pilot Study in Patients With Inflammatory Bowel Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Suboptimal accrual
Sponsor: Entrinsic Bioscience Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2017P000097
Record Dates: First submitted 2018-02-20; First posted 2018-03-01 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Inflammatory Bowel Diseases; Short Bowel Syndrome; Ileostomy - Stoma
MeSH Terms: conditions — Inflammatory Bowel Diseases; Short Bowel Syndrome | interventions — gatorade

STUDY DESIGN:
Intervention Model Description: 4 week randomized into 2 arms, followed by 4 weeks of open label non-randomized follow-up.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Single (physician) blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- amino acid mixture beverage (Experimental): amino acid based hydration beverage. It will be given 8 oz, twice daily for the first 4 weeks of randomized blinded intervention. It will be given in same dose during 4 week open label intervention.
  Interventions: Other: amino acid mixture beverage
- glucose based sports drink (Active Comparator): glucose based hydration beverage. It will be given 8oz, twice daily for the first 4 weeks of randomized blinded intervention.
  Interventions: Other: glucose-based sports drink

INTERVENTIONS:
Other: amino acid mixture beverage — commercially available amino acid mixture. Contains 5 amino acids, electrolytes and natural flavoring.
  Other Names: enterade
  Arms: amino acid mixture beverage
Other: glucose-based sports drink — Commercially available glucose-based sports drink, contains electrolytes, sugar and artificial flavoring.
  Other Names: Gatorade
  Arms: glucose based sports drink

SUMMARY:
This pilot study will examine the benefit of this amino acid based hydration solution in patients with IBD who have undergone a total colectomy and have either ileostomies or jpouches. Findings from this study and possible future studies could have broad implications for patients with malabsorption resulting from many underlying conditions, including IBD.

DETAILED DESCRIPTION:
This pilot study will examine the benefit of this amino acid based hydration solution in patients with IBD who have undergone a total colectomy and have either ileostomies or jpouches. Findings from this study and possible future studies could have broad implications for patients with malabsorption resulting from many underlying conditions, including IBD.

ELIGIBILITY:
Inclusion Criteria:

1. Colectomy with ileostomy

   a. Ileostomy alone with less than 30 cm of small bowel resected i. A diverting ileostomy is permitted
2. Stable disease activity with no or mild inflammation felt not to significantly impact gastrointestinal (GI) output.
3. Any of the following:

   1. Need for IV fluids >2x/month
   2. Intake of > 1.5 liters of oral fluid daily
4. GI output of > 1.3 liters in a 24-hour period for three days each week during a 14 day screening period (does not need to be consecutive days)
5. Stable doses of anti-diarrheal agents, octreotide or Gattex
6. Stable doses of anti-inflammatory agents and/or antibiotics
7. Willing to comply with study visits and assessments, including product intake.

Exclusion:

1. Chronic renal insufficiency glomerular filtration rate (GFR) < 40
2. Significant chronic liver disease altering fluid balance
3. Uncontrolled flare of inflammatory disease

   a. (Inflammation can be present but at a stable at least partly controlled level) b. An anticipated change in medication in the next 3 months i. May be included 8 weeks after changing medications if they are stable c. Anticipated gastrointestinal surgery in the subsequent 3 months i. May be included if they are 4 months out from surgery and stable
4. Diabetes
5. Use of Lactulose/Mannitol solution is contraindicated
6. Current Diagnosis of Cancer

   a. May be included if they are 4 or more months out from cancer therapy (i.e. chemotherapy, etc.)
7. Aversion to the taste of enterade® or inability to take the product as instructed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
GI output | total 8 weeks
  Change in GI output over a 24 hour period as the average of the 3 days every week for two different periods of 4 weeks

SECONDARY OUTCOMES:
Fluid Balance | 8 weeks
  Fluid balance - intake vs output
Tolerability of Drink | 8 weeks
  Taste perception Survey
Quality of Life Index | 8 weeks
  Inflammatory Bowel Disease Questionnaire (IBDQ)
Quality of Life Index | 8 weeks
  SF-36 Questionnaire
Changes in Blood | 8 weeks
  mm Hg
Changes in heart rate | 8 weeks
  Beats per minute
Changes in Lactulose-Mannitol Test | 8 weeks
  The standard test for leaky gut syndrome
Immune Response based on Cytokine Levels | 8 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Brighan and Women's Hospital, Boston, Massachusetts
  - Dartmouth-Hitchcock, Nashua, New Hampshire
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No